CLINICAL TRIAL: NCT01111617
Title: Applications of Realtime fMRI Phase II
Brief Title: Applications of Realtime Functional Magnetic Resonance Imaging (fMRI )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SU-11062007-809; 95194
Record Dates: First submitted 2010-01-29; First posted 2010-04-27 (Estimated); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

ARMS (1):
- Real-Time fMRI (Experimental): Real-Time fMRI
  Interventions: Procedure: Real-time fMRI feedback

INTERVENTIONS:
Procedure: Real-time fMRI feedback — Patients receive real-time fMRI biofeedback to modulate pain

SUMMARY:
The goal of this research program is to determine the potential effectiveness of real-time fMRI training in improving mental control over pain.

DETAILED DESCRIPTION:
A research study that looks at pain and how you experience pain. This research project aims to use virtual reality-based real-time functional Magnetic Resonance Imaging (rtfMRI) to assess brain activation during the experience of pain and while subjects attempt to mentally control their pain response.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Chronic Pain patient or healthy control
* Ability to perform the experimental task

Exclusion Criteria:

* MRI contraindication (metal implants, claustrophobia, pregnant or planning to become pregnant)
* History of psychiatric disorder (at the discretion of the investigator as to whether it interferes with the experimental task)
* History of Blistering

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-01; Primary Completion 2023-11 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
Pain reduction as measured by visual analog scale (VAS) pain report | Within the 2 hour feedback session

SECONDARY OUTCOMES:
Control of brain activity as measured by fMRI analysis | Within the 2 hour feedback session

CONTACTS AND LOCATIONS:
Overall Officials: Sean Mackey, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States